CLINICAL TRIAL: NCT03784404
Title: Trans-vaginal Aspiration With or Without Injection of Surgicel for Treatment of Small Ovarian Endometrioma Before ICSI Cycles. A Randomized Controlled Trial
Brief Title: Trans-vaginal Aspiration of Small Ovarian Endometrioma. Comparison of Two Different Techniques Before ICSI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 45
Record Dates: First submitted 2018-12-20; First posted 2018-12-21 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Ovarian Endometrioma
MeSH Terms: conditions — Endometriosis | interventions — Surgicel; Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non surgicel group (Active Comparator): under sedation transvaginal insertion of spinal needle through the cul de sac under ultrasonographic guidance to reach cyst cavity followed by aspiration of the chocolate material followed by irrigation of the cyst cavity with normal saline solution till complete elimination of the chocolate material
  Interventions: Procedure: Transvaginal aspiration; Drug: Intracytoplasmic sperm injection
- Surgicel group (Active Comparator): under sedation transvaginal insertion of spinal needle through the cul de sac under ultrasonographic guidance to reach cyst cavity followed by aspiration of the chocolate material followed by irrigation of the cyst cavity with normal saline solution till complete elimination of the chocolate material follwed by insertion of 3-4 pieces of small surgicel inside the cyst cavity
  Interventions: Procedure: transvaginal aspiration and surgicel injection; Drug: Intracytoplasmic sperm injection

INTERVENTIONS:
Procedure: Transvaginal aspiration — under sedation transvaginal insertion of spinal needle through the cul de sac under ultrasonographic guidance to reach cyst cavity followed by aspiration of the chocolate material followed by irrigation of the cyst cavity with normal saline solution till complete elimination of the chocolate material
  Arms: Non surgicel group
Procedure: transvaginal aspiration and surgicel injection — under sedation transvaginal insertion of spinal needle through the cul de sac under ultrasonographic guidance to reach cyst cavity followed by aspiration of the chocolate material followed by irrigation of the cyst cavity with normal saline solution till complete elimination of the chocolate material follwed by insertion of 3-4 pieces of small surgicel inside the cyst cavity
  Arms: Surgicel group
Drug: Intracytoplasmic sperm injection — Candidates for the standard long protocol received triptorelin 0.1 mg Subcutanous daily starting from day 21 of the previous cycle. On the second day of the stimulation cycle, pituitary downregulation was confirmed. Controlled ovarian stimulation was then started on day 3 using Human Menopausal Gonadotropin (Menogon; Ferring). The dose of gonadotropin was individualized. The patients were monitored with serial ultrasound and serum E2. When at least 3 follicles reached 18 mm, ovulation was triggered using Human Chorionic Gonadotropin 10000 IU (Epifasi 10000 IU; Eipico, Tenth of Ramadan, Egypt) IM and ovum pickup was performed 35 hours later.
  All cases received luteal support in the form of progesterone 400 mg twice daily. Embryo transfer was done on day 3 or 5 using Labotect semi-rigid catheter (Labotect GmbH, Kassel area, Germany) under abdominal ultrasound guidance.

SUMMARY:
women candidate for ICSI and having ovarian endometrioma smaller than 5 cm will be randomized to either transvaginal aspiration alone or transvaginal aspiration follwed by injection of small parts of oxidized regenerated cellulose within the cyst cavity during the cycle that preceded the induction cycle of ICSI

DETAILED DESCRIPTION:
women candidate for ICSI and having ovarian endometrioma smaller than 5 cm will be randomized to either transvaginal aspiration alone or transvaginal aspiration follwed by injection of small parts of oxidized regenerated cellulose within the cyst cavity during the cycle that preceded the induction cycle of ICSI.

Transvaginal aspiration will be done under ultrasonographic guidance with spinal needle insertion inside the cyst cavity followed by aspiration of the chocolate material from the cyst & then irrigation of the cyst cavity with normal saline solution till complete elimination of the chocolate material. The needle will be withdrawn in women in non-Surgicel group while injection of small pieces of surgicel inside the cyst cavity will be done for women in the surgicel group followed by withdrawal of the needle.

ELIGIBILITY:
Inclusion Criteria:

* Subfertile women indicated for ICSI
* having a single endometrioma of less than 5 cm with typical sonographic criteria; a cyst with 1 to 4 locules and ground glass appearance of the cyst fluid with no papillary projections and no or minimal vascularization of the cyst capsule. Since endometriotic cysts measuringmore than 1 cm are readily diagnosed by ultrasound,25 we chose a diameter of 2 cm as the lower limit to declare a cyst as endometrioma.
* All cases had a normal uterine cavity demonstrated by ultrasonography and hysteroscopy.

Exclusion Criteria:

* bilateral or multiple endometriomas, lesions of more than 5 cm or showing atypical sonographic features presence of uterine pathology (eg, polyp or fibroid)
* follicle-stimulating hormone (FSH) of more than 10,
* body mass index of more than 30, age more than 40 years,
* cases who received previous GnRH therapy for treatment of endometriosis within 12 months of the study
* patients who received oral contraceptive pills or any form of hormones for the previous 3 months,
* patients with previous surgical resection of endometrioma
* severe male factor.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 14 days after embryo transfer
  documentation of intrauterine fetal sac using transvaginal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided